CLINICAL TRIAL: NCT06768567
Title: Evaluation of Effect of Hemostasis Time on Partial Pulpotomy in Mature Permanent Teeth With Clinical Signs Indicative of Irreversible Pulpitis
Brief Title: Evaluation of Hemostasis Time on Partial Pulpotomy in Teeth With Clinical Signs Indicative of Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vinita yadav
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Irreversible Pulpitis; Partial Pulpotomy
Keywords: partial pulpotomy; hemostatsis time

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemostasis time upto 6 minutes (Active Comparator): after partial pulpotomy, procedure pulp wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 minutes and will be repeated if required and time taken to achieve hemostasis will be recorded using stop watch.
  Interventions: Procedure: effect of hemostasis time on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.
- hemostasis time 7 to 12 minutes (Experimental): after partial pulpotomy, procedure pulp wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 minutes and will be repeated if required and time taken to achieve hemostasis will be recorded using stop watch.Root canal therapy will be initiated in cases in which haemostasis is not achieved even after 12 minutes.
  Interventions: Procedure: effect of hemostasis time on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

INTERVENTIONS:
Procedure: effect of hemostasis time on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis. — After caries removal and pulp exposure pulp tissue is amputated and pulpal wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 to 3 minutes and will be repeated if required and time taken to achieve hemostasis will be recorded using stop watch. Teeth in which bleeding will be controlled within 6 mins will be placed in Group A, while those in which it gets controlled between 7 to 12 mins will be included in Group B. Root canal therapy will be initiated in cases in which haemostasis is not achieved even after 12 minutes. Followed by capping with 2-3mm layer of MTA. A layer of RMGIC will be placed over the MTA. Then the tooth will be permanently restored with composite resin.

SUMMARY:
The aim of this prospective study is to investigate the influence of time taken to achieve hemostasis on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

OBJECTIVE:-

1. To evaluate clinical and radiographic success of time taken to achieve hemostasis on outcome of partial pulpotomy in mature permanent teeth with clinical signs indicative of irreversible pulpitis.
2. To evaluate OHRQoL and pain incidence & severity after partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

Participants will of age group 18 to 45 years will be included and divided into two groups based on hemostasis time:

I(Intervention) - 6minutes C (Comparison) - 7-12 minutes

DETAILED DESCRIPTION:
TITLE:- Evaluation of hemostasis time on partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

P (Population) - Mature permanent molars with clinical signs of irreversible pulpitis.

I (Intervention) - 6minutes C (Comparison) - 7-12 minutes O (Outcome) - Assessment of clinical and radiographic success at 12 months of follow up .

Assessment of OHRQoL at baseline, post-operatively every 24 hours for 1 week & incidence and severity of pain at baseline and post-operatively every 24 hours till 1 week.

Time taken to achieve hemostasis has been suggested as a reliable surrogate measure to determine the depth of inflammation in the pulp. In absence of any other intraoperative indicator, it serves as a useful guide to the extent of pulp tissue removal required during pulpotomy. This trial will help formulate evidence based guideline regarding time for hemostasis advisable to achieve optimum success during pulpotomy in teeth with signs indicative of irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent mandibular molars with carious pulp exposures and signs suggestive of irreversible pulpitis.
* vital pulp with demonstrable bleeding upon entry.
* The tooth is restorable.
* Tooth with mobility and probing depth within normal limits.
* Soft tissues around the tooth are normal with no swelling or sinus tract.
* No evidence of chronic apical periodontitis (PAI 1,2)

Exclusion Criteria:

* patients who report history of antibiotic intake in past 1 month or analgesic intake in past 3 days.
* pregnant women.
* absence of opposing teeth
* 3rd molars
* medically compromised patients .
* Tenderness on percussion positive
* pathologic mobility

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
1.Clinical success rate | baseline to 12 months
  Clinical criteria of success:-
  1. No pain or discomfort except for the first few days after treatment.
  2. No tenderness to palpation or percussion and the tooth is functional.
  3. Normal mobility and probing pocket depth.
  4. Healthy soft tissues around teeth with no swelling, sinus tract.
2.Radiographic success rate | baseline to 12 months
  Radiographic success criteria:-
  1. No pathosis such as root resorption, furcal pathosis or new periapical pathosis evident on the radiograph.
  2. Complete radiographic healing

SECONDARY OUTCOMES:
Post Operative Pain | Baseline to 7 days]
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain
OHRQoL assessment | baseline and at 24 hours, day 2, day 3, day4, day 5, day 6 and day 7 after the treatment.
  OHIP-14 questionnare will be used to assess the quality of life.It consists of questionnaire in seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. It will be scored using a Lickert scale:
  never=0; hardly ever=1; occasionally=2; fairly often=3; very often=4. Total score will be calculated ranging from 0-56, with higher score denoting the worst OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pankaj Sangwan, MDS, Study Director — PGIDS, Rohtak, Haryana 124001
Locations (1):
- PGIDS, Rohtak, Haryana, India